CLINICAL TRIAL: NCT04228029
Title: Does Carboxytherapy Play a Role in Alopecia Areata Either Solely or in Combination? Comparative Study for Treatment of Alopecia Areata Using Carboxytherapy and Intralesional Steroids
Brief Title: Comparative Study for Treatment of Alopecia Areata Using Carboxytherapy and Intralesional Steroids
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Rana F Hilal, MD, Lecturer of dermatology, faculty of Medicine, Cairo University., Kasr El Aini Hospital
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: KasrEliniH
Record Dates: First submitted 2020-01-08; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Carboxytherapy (Active Comparator)
  Interventions: Device: Carboxytherapy
- Intralesional steroids (Active Comparator)
  Interventions: Drug: Intralesional Steroid Injection
- Combination of carboxytherapy and intralesional steroids (Active Comparator)
  Interventions: Device: Carboxytherapy; Drug: Intralesional Steroid Injection

INTERVENTIONS:
Device: Carboxytherapy — Carbon dioxide (CO2) gas in injection form
  Arms: Carboxytherapy; Combination of carboxytherapy and intralesional steroids
Drug: Intralesional Steroid Injection — triamcinolone acetonide 8 mg/mL
  Arms: Combination of carboxytherapy and intralesional steroids; Intralesional steroids

SUMMARY:
Patients with three lesions of alopecia areata are randomly recruited in this study. Each lesion is randomized in to receiving either carboxytherapy in one lesion, intralesional steroids in another lesion and combination of both in the third lesion.

Treatment period is 3 months followed by a follow-up period of 2 months.

ELIGIBILITY:
Inclusion Criteria:

* early localized scalp alopecia areata
* patients who did not receive any medication for at least 2 months before starting the study Patients who agreed to join the study and signed written consent.

Exclusion Criteria:

* pregnant, and lactating females and those with unrealistic expectation.
* Alopecia totalis or universalis or ophiasis or cicatrising alopecia
* Usage of systemic treatment of alopecia areata 2 months prior to the study.
* Any scalp lesion within the treated area
* Bleeding diathesis, severe anemia or platelet disorders
* Medical conditions such as autoimmune diseases.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2020-02-20 (Estimated); Study Completion 2020-04-20 (Estimated)

PRIMARY OUTCOMES:
Severity of Alopecia Tool (SALT) score | 6months-1 year
  evaluate efficacy of carboxytherapy versus intralesional steroids versus combination of both Minimum value is 0% and maximum value is100% the higher the score the more the hair loss
Dermoscopy | 6months-1 year
  evaluate efficacy of carboxytherapy versus intralesional steroids versus combination of both through counting number dystrophic hair, tapered hair, regrowing hair, black dots, and yellow dots
blinded observer evaluation by use of photography | 6months-1 year
  evaluate efficacy of carboxytherapy versus intralesional steroids versus combination of both
patient satisfaction rate | 6months-1 year
  evaluate efficacy of carboxytherapy versus intralesional steroids versus combination of both

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr ElAiny Hospital, Cairo university, Cairo, El Manial, Egypt

REFERENCES:
- [Derived] Metwally D, Abdel-Fattah R, Hilal RF. Comparative study for treatment of alopecia areata using carboxy therapy, intralesional corticosteroids, and a combination of both. Arch Dermatol Res. 2022 Mar;314(2):167-182. doi: 10.1007/s00403-021-02201-6. Epub 2021 Mar 19. PMID 33742252